CLINICAL TRIAL: NCT02807805
Title: A Phase II Study With a Lead-in Safety Phase of Abiraterone in Combination With PDMX1001/Niclosamide in Castration-Resistant Prostate Cancer (CRPC)
Brief Title: Abiraterone Acetate, Niclosamide, and Prednisone in Treating Patients With Hormone-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mamta Parikh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Mamta Parikh, Associate Professor, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 871875; UCDCC#260 (Other: UC Davis IRB); UCDCC#260 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH); NCI-2016-00779 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-06-13; First posted 2016-06-21 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Prostate Carcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer
Keywords: castration resistant prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Niclosamide; Prednisone; deltacortene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (abiraterone acetate, niclosamide, prednisone) (Experimental): Patients receive abiraterone acetate PO QD, niclosamide PO BID and prednisone PO BID. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abiraterone Acetate; Drug: Niclosamide; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Zytiga
Drug: Niclosamide — Given PO
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone

SUMMARY:
This phase II trial studies the side effects and how well abiraterone acetate, niclosamide, and prednisone work in treating patients with hormone-resistant prostate cancer. Androgens can cause the growth of prostate cells. Hormone therapy using abiraterone acetate may fight prostate cancer by lowering the amount of androgen the body makes. Niclosamide is a drug that may block another signal that can cause prostate cancer cell growth. Prednisone is a drug that can help lessen inflammation. Giving abiraterone acetate, niclosamide, and prednisone may be a better treatment for patients with hormone-resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the prostate-specific antigen (PSA) response that is a 50% or more reduction from the baseline.

SECONDARY OBJECTIVES:

I. To determine the overall response as determined by the Prostate Cancer Working Group 2 criteria (PCWG2).

II. To evaluate the progression-free survival (PFS) and overall survival of CRPC patients treated with PDMX1001/niclosamide (niclosamide), abiraterone (abiraterone acetate) and prednisone.

III. To assess the toxicity of PDMX1001/niclosamide, abiraterone and prednisone given in combination.

OUTLINE:

Patients receive abiraterone acetate orally (PO) once a day (QD), niclosamide PO twice a day (BID) and prednisone PO BID. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed cancer of prostate (CaP); CaP can be recurrent disease after definitive therapy (radical prostatectomy or radiation therapy) for localized CaP, or metastatic CaP
* Patients must have CaP deemed to be castration-resistant by one or more of the following criteria (despite androgen deprivation when applicable):

  * Progression of unidimensionally measurable disease assessed within 42 days prior to initial administration of drug
  * Progression of evaluable but not measurable disease assessed within 42 days prior to initial administration of drug for PSA evaluation and for imaging studies (e.g, bone scans)
  * Rising PSA, defined as at least two consecutive rises in PSA to be documented over a reference value (measure 1); the first rising PSA (measure 2) should be taken at least 7 days after the reference value; a third confirmatory PSA measure (second [2nd] beyond the reference level) should be greater than the second measure, and it must be obtained at least 7 days after the 2nd measure; if this is not the case, a fourth PSA measurement is required to be taken and be greater than the second measure
* Measurable disease is not required

  * Patients who have measurable disease must have had X-rays, scans or physical examinations used for tumor measurement completed within 28 days prior to initial administration of drug
  * Patients must have non-measurable disease (such as nuclear medicine bone scans) and non-target lesions (such as PSA level) assessed within 28 days prior to initial administration of drug
  * Soft tissue disease that has been radiated within two months prior to registration is not assessable as measurable disease; soft tissue disease that has been radiated two or more months prior to registration is assessable as measurable disease provided that the lesion has progressed following radiation; as the biology of previously irradiated tumors may be different from non-irradiated tumors, patients must have at least one measurable lesion outside the previously irradiated region in order to be considered to have measurable disease
  * If PSA is the only indicator of disease and patients do not have any metastatic disease, PSA value must be 5.0 or higher
* Patients must have been surgically or medically castrated; if the method of castration was luteinizing hormone-releasing hormone (LHRH) agonists (leuprolide or goserelin) or antagonists (degarelix), then the patient must be willing to continue the use of LHRH agonists or antagonists; serum testosterone must be at castration levels (< 50 ng/dL) within 3 months prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 6 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 1.5 × institutional upper limit of normal
* Creatinine =< 1.5 x institutional upper limit of normal
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of abiraterone and PDMX1001/niclosamide administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents within the preceding 4 weeks
* Patients on herbs or other alternative medicines for the treatment of prostate cancer, including but not limited to saw palmetto, PC-SPES
* Patient has received abiraterone or ketoconazole for the treatment of prostate cancer; however, previous treatment with other hormonal therapy (bicalutamide, enzalutamide, flutamide and nilutamide) or chemotherapy (docetaxel, cabazitaxel or mitoxantrone) is allowed
* Other malignancies within the past 3 years except for adequately treated basal or squamous cell carcinomas of the skin or other stage 0 or I cancers
* Patients with known brain metastases should be excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to abiraterone or PDMX1001/niclosamide
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active bleeding diathesis
* History of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol
* Patients with symptomatic metastatic prostate cancer such as moderate to severe pain, impaired organ function or spinal cord compression will be excluded from this study unless these issues have been taken care of

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-10; Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
PSA response rate | Up to 2 years
  Percent of patients achieving greater than or equal to 50% PSA declines following initiation of treatment

SECONDARY OUTCOMES:
Incidence of dose limiting toxicity defined as any grade III non-hematologic toxicity not reversible to grade II or less within 96 hours, or any grade IV toxicity | 4 weeks
  Graded according to National Cancer Institute Common Terminology Criteria for Adverse Events 4.0. Adverse events and adverse events of grade 3 or higher will be listed for each patient and summarized by body system in a frequency table.
Overall response as determined by PCWG2 criteria | From the time measurement criteria are met for complete response/partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 2 years
Overall survival | Up to 2 years
  Will be estimated using the product-limit method of Kaplan and Meier; medians and 95% confidence intervals will be computed.
PFS | Up to 2 years
  Will be estimated using the product-limit method of Kaplan and Meier; medians and 95% confidence intervals will be computed. Will be compared with the historic control of abiraterone alone.

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Parikh, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States